CLINICAL TRIAL: NCT06660771
Title: Polygraphic Evaluation of the Effects of Functional Orthodontic Treatment with Twin Block and Herbst Appliances on Sleep Quality: a Randomized Clinical Trial
Brief Title: Evaluation of Functional Orthodontic Treatment on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gökçenur Gökçe Kara (Other)
Collaborators: Izmir Katip Celebi University (Other); Ege University (Other)
Responsible Party: Sponsor-Investigator, Gökçenur Gökçe Kara, ASSOCIATE PROFESSOR, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-07

CONDITIONS: Sleep Apnea Syndromes in Children; Functional Orthodontic Treatment; Mandibular Retrognathia; Upper Airway
Keywords: Obstructive sleep apnea; Herbst; Twin Block
MeSH Terms: conditions — Micrognathism; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: 2-arm parallel trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Herbst (Experimental): The Herbst appliance is fixed and rigid functional appliance. It consists of attachments (casted splints) in the lateral segments of both jaws which are connected by a telescoping mechanism from the upper posterior to the lower anterior region resulting in mandibular bite jumping.
  Interventions: Procedure: Functional orthodontic treatment
- Twin Block (Experimental): Twin-block appliance is used with two separate acrylic plates for the lower and upper jaw.
  It consists of acrylic bite blocks that lock together at a 70° angle, allowing the mandible to be positioned in front.
  Interventions: Procedure: Functional orthodontic treatment

INTERVENTIONS:
Procedure: Functional orthodontic treatment — The patients were treated with Twin block and Herbst functional appliances. Alginate impressions and a protrusive wax bite were taken for the construction of each appliance. Each device was fitted and then reviewed 4-6 weeks later. First group was treated with Twin block which was manufactured basically according to the original design described by Clark. The overjet was measured from the patients in centric relationship and maximum protrusion position, and construction bite was recorded with 70% of the total advancement capacity of the mandible and 2-4 mm above the freeway space vertically. Overjet measurements were made at each session and active treatment was terminated when a normal overjet in the retracted position was recorded.
  Second group was treated with the stainless-steel crown Herbst appliance, included crowned maxillary first molars and mandibular first premolars. The construction bite was recorded with the mandible forward by edge-to-edge incisor position.

SUMMARY:
Functional appliances are used in the treatment of Class II anomalies caused by mandibular rethrognathia. Herbst which is a fixed and rigid functional appliance and TWB which is removable appliance can be successful in the treatment of mandibular retrognathia in a short period of six to eight months during the pubertal growth phase. An increase in the upper airway size occurs as a result of functional orthopedic treatment devices eliminating the problem of mandibular retrognathia and stimulating mandibular growth. The aim of this randomized controlled trial was to evaluate the effects of TWB and Herbst appliances on sleep quality in children with obstructive sleep apnea. The null hypothesis was that there is no difference for the sleep quality between the appliances.

DETAILED DESCRIPTION:
Introduction: This multicenter clinical study aimed to investigate the effects of twin block (TB) and Herbst functional appliances on sleep quality in children with OSAS and mandibular retrognathia. Methods: A total of 46 patients having mandibular retrognathia and identified with OSA were divided randomly into two groups: twin block (TB) and Herbst functional appliances. Changes in sleep parameters at baseline and an avarage of 8-month follow-up detected by polygraphy and Pittsburg Sleep Quality Index (PSQI) were the primary outcome. Treatment of the mandibular retrognathia was the secondary outcome. hapiro Wilk test and Q-Q graphs were used to examine the distribution assumptions of continuous variables according to groups. Mann Whitney U test was used to evaluate two independent group means or distributions of continuous measurements. Paired sample t test or Wilcoxon signed rank test was used to evaluate the differences between the baseline and follow-up times at p < 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* no prior orthodontic treatment, nasal, tonsillar, or adenoid surgery
* absence of any oral, nasal or systemic disease
* the existence of skeletal Class II and dental Class II Division 1 malocclusion (ANB >4°; SNB <80°; incisor overjet >3 mm)
* requiring functional orthodontic treatment
* Individuals are in the MP3cap and S period according to hand-wrist films, and in the CS3 and CS4 period using the CVM method
* patients with OSA (apnea/hypopnea index (AHI)>1/h

Exclusion Criteria:

* body mass index (BMI) ≥ 30 (weight (kg)/height (m2))
* the presence of nasopharyngeal pathologies, craniofacial anomalies, , systemic disorder, or weak oral hygiene
* history of previous orthodontic treatment

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Correction of mandibular retrognathia | Following 6-8 months active treatment
  A normal or corrected overjet in the retracted position

SECONDARY OUTCOMES:
Polygraphic assessment of sleep parameters | Following 6-8 months active treatment
  Changes in apnea hypopnea index (AHI)
Polygraphic assessment of sleep parameters | Following 6-8 months active treatment
  Changes in number of apnea and hypopnea
Polygraphic assessment of sleep parameters | Following 6-8 months active treatment
  Changes in number of hypopnea
Polygraphic assessment of sleep parameters | Following 6-8 months active treatment
  Changes in desaturation index
Polygraphic assessment of sleep parameters | Following 6-8 months active treatment
  Changes in lowest desaturation
Polygraphic assessment of sleep parameters | Following 6-8 months active treatment
  Changes in average saturation
Polygraphic assessment of sleep parameters | Following 6-8 months active treatment
  Changes in the value of Supin AHI

CONTACTS AND LOCATIONS:
Overall Officials: Gökçenur Gökçe Kara, Principal Investigator — Marmara University
Locations (1):
- Gökçenur Gökçe Kara, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided